CLINICAL TRIAL: NCT01164241
Title: Natural History of Severe Allergic Inflammation and Reactions
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100148; 10-I-0148
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-10-22

CONDITIONS: PGM3 Deficiency; Eosinophilic and/or Atopic Dermatitis; OSMR Deficiency; Primary Localized Cutaneous Amyloidosis; Hereditary Alpha-tryptasemia
Keywords: Tryptase; Dermatitis; Eosinophilia; Anaphylaxis; Natural History; Genetics
MeSH Terms: conditions — Amyloidosis, Primary Cutaneous; Hereditary alpha-tryptasemia syndrome; Dermatitis; Eosinophilia; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Eczema
- 2: unaffected relatives
- 3: healthy volunteers
- 4: other allergic phenotypes

SUMMARY:
Background:

- Allergic inflammation is central to allergy-related diseases and disorders, such as asthma, food allergies, and atopic dermatitis. Atopic dermatitis, commonly called eczema is a chronic, noncontagious skin condition, usually starting in the first years of life, which causes itching and scaling of an individual s skin. Because atopic dermatitis is a common condition in children who have allergy-related diseases, including asthma, researchers are interested in studying both individuals with atopic dermatitis and their close relatives (parents and children) to better understand how allergy-related diseases develop and progress. In addition, some patients with inherited disorders with features including atopic dermatitis or other aspects of allergy such as food allergy, asthma, hay fever, hives, and others, will also be seen.

Objectives:

- To study the natural history of diseases of allergic inflammation, such as atopic dermatitis or genetic disorders associated with allergic inflammation.

Eligibility:

* Children and adolescents between 1 month and 21 years of age who have a documented history of moderate to severe atopic dermatitis.
* Individuals between 1 month and 80 years of age who have a suspected genetic or inherited allergy disorder related to atopic dermatitis or allergic pathways.
* Child and adult relatives of eligible participants will also be studied on this protocol.

Design:

* The study will require one initial visit to the National Institutes of Health Clinical Center (lasting 1-5 days), as well as any required follow-up visits for treatment and research studies. Participants will receive treatment for atopic dermatitis and other allergic diseases as part of the study for up to 1 year.
* Participants will have some or all of the following tests as part of this study:
* A detailed physical examination and medical history
* Allergy skin prick testing to examine participants' responses to different allergens.
* Blood samples for additional allergen testing, testing the immune system, and other research purposes
* Skin punch biopsy to take a skin sample
* Lung function tests to measure airflow from the lungs and inflammation
* Food-related tests to diagnose potential food allergies
* Leukapheresis to collect white blood cells only
* Research samples, including stool specimens, saliva samples, buccal swabs (to collect cells from the inside of the cheek), and skin cell samples
* Clinical digital photography to provide images of affected and healthy skin.
* Participants will be asked to return for follow-up visits and tests for up to 1 year after the initial visit(s).

DETAILED DESCRIPTION:
Background:

Allergic inflammation is central to the pathogenesis of allergic diseases, including atopic dermatitis, asthma, allergic rhinitis, and food allergy. These disorders are common, affecting up to 50 million Americans, and their pathophysiology remains poorly understood. Among allergic diseases, atopic dermatitis is common, with a prevalence of up to 20% in children. It is associated with the most dramatic elevations of IgE levels and most prominent T-helper type 2 cell (Th2) inflammation, and treatment remains challenging. Atopic dermatitis, eosinophilic inflammation, and systemic immediate hypersensitivity reactions are heralding manifestation of allergic disease in many children, making these ideal disorders for studying the effector mechanisms promoting the development and progression of allergic diseases. In addition to these manifestations, there are also a number of characterized genetic and congenital diseases, most presenting in childhood, that have prominent allergic manifestations, including dermatitis, or affect atopic pathways. These disorders provide further opportunity for advancing our understanding of the genetics and pathophysiology of diseases of allergic inflammation. The NIAID Laboratory of Allergic Diseases (LAD) has a long interest in exploring the mechanisms of allergic inflammation. Utilizing the resources of the LAD and the NIH Clinical Center, we will advance our understanding of allergic inflammation and the genetics and pathogenesis of allergic diseases through the study of these patients. The findings of this protocol will have implications for improved diagnosis, treatment and prevention of allergic diseases, including atopic asthma.

Objectives:

The overall goal of this exploratory protocol is to study the natural history of individuals with severe allergic inflammation and hypersensitivity reactions, focusing on individuals and families with known or suspected inherited or acquired genetic causes for these clinical manifestations. Research studies obtained from blood, skin, saliva, bone marrow, and other tests obtained from participants will be used to explore the genetic, immunologic, structural, and microbiologic abnormalities of these diseases. Research studies obtained from blood samples, allergy skin testing, and skin biopsies of unaffected relatives and healthy volunteers will be used as controls for assays and genetic tests. Results of research studies will be correlated with clinical features of allergic manifestations of disease and response to therapy.

Eligibility:

Subjects eligible for enrollment in this study include children and a subset of adults with a known or suspected inherited or acquired genetic allergic disorder leading to severe allergic inflammation or reactions. Unaffected relatives of an enrolled subject (both children and adults) and healthy adult volunteers will also be eligible for separate enrollment.

Design:

The initial enrollment for this protocol will be 1500 primary subjects. In addition, approximately 500 healthy or affected parents, siblings, or other relatives may be enrolled for initial history and clinical and research laboratory evaluation only. Approximately 150 unrelated healthy adult volunteers will also be enrolled. Affected subjects in this study will receive standard care for allergic diseases, both outpatient and inpatient, during the period of enrollment and will receive extensive evaluation as clinically indicated, in addition to research studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subject or unaffected relatives must:

  1. Be at least 2 years of age and less than or equal to 21 years of age at the time of enrollment and have documented history of severe allergic inflammation or hypersensitivity, that began in the first 5 years of life, that is moderate to severe, and with continued inflammation or

     recurrent flares in the preceding 3 months. Patients greater than 21 years of age with a history of disease in the first 5 years of life and/or, if in the opinion of the PI or AIs, the patient would be of interest to fulfill the objectives of the study.

     OR
  2. Be 2-80 years of age with a known or suspected genetic or congenital disorder associated with severe allergic inflammation or

     hypersensitivity, as determined by the PI or AIs.

     OR
  3. Be an a relative of a patient enrolled in the protocol.
* Have a private physician to provide local continuity of care.
* Provide a letter of referral, with copies of pertinent medical history and laboratory studies as indicated, from the prospective study participant s referring physician; this is not a requirement for healthy relatives.
* Be willing to donate blood, buccal swabs, saliva, skin and nasal swabs for research and clinical studies and for storage to be used for future research and genetic testing; for unaffected relatives, be willing to donate blood and/or undergo allergy skin testing, in addition to having blood samples stored for future research and genetic testing.
* Pregnant women or women who become pregnant are eligible to participate or continue participation on the study.

Healthy Volunteer must:

* Be at least 18 years old and no greater than 80 years old, and able to provide informed consent.

  2. Have no history of severe or recurrent allergic diseases or reactions.
* Be willing to have samples stored for research and genetic testing.

EXCLUSION CRITERIA:

Any subject with any of the following criteria will be excluded:

* Presence of conditions that, in the judgment of the investigator or the referring physician, may put the subject at undue risk or make them unsuitable for participation in the study.
* Inability or refusal to undergo study procedures.
* Inability to participate for the duration of the study.

Any unaffected relative or healthy volunteer with any of the following criteria will be excluded:

* Presence of conditions that, in the judgment of the investigator or the referring physician, may put the subject at undue risk or make them unsuitable for participation in the study.
* Inability or refusal to undergo study procedures.
* Inability to provide informed consent.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Referrals for severe, familial or atypical allergic disease from throughout the country and world-- either physician or self referrals.
Sampling Method: Non-Probability Sample
Enrollment: 945 (Actual)
Dates: Start 2010-07-12 (Actual)

PRIMARY OUTCOMES:
SCORAD | At initial and single follow up visit 1-2 months after.
  Severity of atopic dermatitis, only taken when present.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela A Guerrerio, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Glover SC, Carter MC, Korosec P, Bonadonna P, Schwartz LB, Milner JD, Caughey GH, Metcalfe DD, Lyons JJ. Clinical relevance of inherited genetic differences in human tryptases: Hereditary alpha-tryptasemia and beyond. Ann Allergy Asthma Immunol. 2021 Dec;127(6):638-647. doi: 10.1016/j.anai.2021.08.009. Epub 2021 Aug 13. PMID 34400315
- [Background] Lyons JJ, Milner JD. Primary atopic disorders. J Exp Med. 2018 Apr 2;215(4):1009-1022. doi: 10.1084/jem.20172306. Epub 2018 Mar 16. PMID 29549114
- [Derived] Lexmond WS, Goettel JA, Lyons JJ, Jacobse J, Deken MM, Lawrence MG, DiMaggio TH, Kotlarz D, Garabedian E, Sackstein P, Nelson CC, Jones N, Stone KD, Candotti F, Rings EH, Thrasher AJ, Milner JD, Snapper SB, Fiebiger E. FOXP3+ Tregs require WASP to restrain Th2-mediated food allergy. J Clin Invest. 2016 Oct 3;126(10):4030-4044. doi: 10.1172/JCI85129. Epub 2016 Sep 19. PMID 27643438
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-I-0148.html